CLINICAL TRIAL: NCT07381959
Title: Biomarkörer för hjärnskada Hos Barn Med hjärntumör
Brief Title: Biomarkers of Brain Injury in Children With Brain Tumors
Acronym: BiomarkCBT
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Region Blekinge (Unknown); Region Dalarna (Unknown); Region Gotland (Unknown); Region Gävleborg (Other); Region Uppsala (Unknown); Region Halland (Other); Region Jämtland Härjedalen (Other); Region Jönköping County (Other Government); Region Kalmar län (Unknown); Region Kronoberg (Unknown); Region Norrbotten (Unknown); Region Skåne (Unknown); Region Stockholm (Other Government); Sormland County Council, Sweden (Other); Region Värmland (Unknown); Region Västerbotten (Other Government); Region Västernorrland (Unknown); Region Västmanland (Other); Region Örebro län (Unknown); Region Östergotland (Unknown); Göteborg University (Other); Västra Götalandsregionen (Other)
Responsible Party: Sponsor
Other Study IDs: LUL-964455
Record Dates: First submitted 2025-12-29; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor; Childhood Cancer; Childhood Brain Tumor
Keywords: Radiotherapy; Cranial radiation therapy; Plasma biomarkers; Extracellular vesicles; Proteomics; Childhood brain tumor
MeSH Terms: conditions — Brain Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA)- and sodium citrate collection tubes will be used to collect plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A - Radiation: Children diagnosed with primary brain tumors who are treated with surgery and radiation therapy, and/or other cancer treatment (n=160).
- Group B - Radiation-naive: Children diagnosed with primary brain tumors who are treated with surgery and/or other cancer treatment, but not radiation therapy (n=200).
- Group C - Healthy Controls: Healthy children without brain tumors (n=200).

SUMMARY:
The goal of this observational study is to identify biomarkers of treatment-induced brain injury in children treated for primary brain tumors. The main question it aims to answer is:

Can investigators identify sensitive plasma biomarker(s) of treatment-induced brain injury in children with primary brain tumors?

Researchers will compare results between different treatment modalities (surgery, chemotherapy, radiation versus radiation-naive) and a healthy age- and sex-matched control population, to identify treatment-specific biomarkers.

Participants will provide plasma samples at the following time points: before surgery, 1-2 weeks after surgery, as well as at 3-, 6-, 12-, 18-, 24-, and 36 months after surgery. Participants who receive radiation treatment will also provide plasma samples before and during treatment (approximately every 2 weeks). Where possible, plasma samples are also collected before the start of any new treatment (e.g., chemotherapy). Healthy controls will provide samples once.

ELIGIBILITY:
Inclusion Criteria, Group A (treated with radiation):

* Age 0-17 years old, AND
* Diagnosed with primary brain tumor through surgery, biopsy, or other diagnostic method (e.g., for germinoma) at Uppsala University Hospital or at another university hospital in Sweden, AND
* Referred for radiotherapy at Skandion Clinic in Uppsala and/or at their local hospital (in some cases), with/without the addition of other cancer treatments.

Inclusion Criteria, Group B (treated without radiation/radiation naive):

* Age 0-17 years old, AND
* Diagnosed with primary brain tumor through surgery, biopsy, or other diagnostic method (e.g., for optic pathway glioma in neurofibromatosis type 1 and germinoma) at Uppsala University Hospital or at another university hospital in Sweden, AND
* Not referred to radiotherapy and treated with/without the addition of other cancer treatments.

Inclusion Criteria, Group C (healthy control group):

* Age 0-17 years old at time of recruitment

Exclusion Criteria, Groups A + B:

* Diagnosed with a tumor only in the spinal cord (solitary spinal tumor).
* Diagnosed with a tumor considered palliative already at diagnosis (e.g., diffuse intrinsic pontine glioma)

Exclusion Criteria, Group C:

* Have diagnosis of chronic disease that requires continuous medication.

Exclusion Criteria, all groups:

* Unable to provide informed consent due to language difficulties.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Groups A and B will be selected from all children, 0-17 years of age, in Sweden with primary (newly diagnosed) brain tumors.
  Group C will be selected from:
  * Healthy sibling controls to other study participants, OR
  * Siblings to other children admitted to Uppsala University Hospital, OR
  * Other healthy children for example those who attend Uppsala University Hospital for another reason (e.g., minor elective daycare surgery).
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker(s) of brain injury | From enrollment until the end of study follow-up (up to 3 years after start of primary behandling for primary brain tumor, such as operation for brain tumor)
  Exploratory. "Brain injury" includes, e.g., changes visible on magnetic resonance imaging and neurocognitive follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Arja Harila, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data can only be shared upon reasonable request, with appropriate approvals in place.